CLINICAL TRIAL: NCT03596359
Title: Effect of Self-care Education With Teach-Back Method on Quality of Life in Heart Failure Patients
Brief Title: Teach-Back Method on Quality of Life in Heart Failure Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baqiyatallah Medical Sciences University (Other)
Responsible Party: Principal Investigator, Mohammad Sadegh Bagheri Baghdasht, Principal Investigator, Baqiyatallah Medical Sciences University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: IR.BMSU.Rec.1394.144
Record Dates: First submitted 2018-06-25; First posted 2018-07-23 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Heart Failure
Keywords: Self Care; Heart Failure; Quality of Life; Teach-Back
MeSH Terms: conditions — Heart Failure | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Self-care behaviors training with Teach-Back method within 15 to 45 minutes was done on the Test group
  Interventions: Behavioral: Education with Teach-Back method
- Control group (Active Comparator): The control group received routine treatment
  Interventions: Other: Received routine treatment

INTERVENTIONS:
Behavioral: Education with Teach-Back method
  Arms: Test group
Other: Received routine treatment
  Arms: Control group

SUMMARY:
This study determines effect of education with Teach-Back method in patients with Heart failure. In this randomized clinical trial, 70 patients with Heart failure hospitalized in year 2016-17 were selected and they were randomly divided into control group and test group.Self-care behaviors training with Teach-Back method within 15 to 45 minutes was done on the case group, and control group received routine treatment. Information have collected whit Demographic questionnaire and SF36 questionnaire before and after training. Data were analyzed by Spss version18 And there were analyzed by descriptive statistics and Chi-square, Independent T-test, Paired T-test and Co-variance tests.

ELIGIBILITY:
Inclusion Criteria:

* Age from 45 to 85
* Heart failure diagnosed six months ago
* The Ejection Fraction less than 45
* Have reading and writing skills
* Have perfect consciousness
* Fluency in Persian

Exclusion Criteria:

* Patient do not cooperate with researchers
* The inability of each sample to continue cooperation during the study because of the problem or acute disease.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-11-18 (Actual); Primary Completion 2017-03-02 (Actual); Study Completion 2017-05-20 (Actual)

PRIMARY OUTCOMES:
SF 36 questionnaire | Up to 48 hours
  SF36 questionnaire was used to measuring the quality of life
Demographic questionnaire | 24 hours
  Demographic questionnaire was used to collect information